CLINICAL TRIAL: NCT04076085
Title: Effect of Unsupported Upper Extremity Exercise Versus Lower Extremity Exercise in Individuals With Chronic Obstructive Disease (COPD) on Dyspnea and Peak Flow Rate
Brief Title: Effect of Extremity Exercise in COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King Khalid University (Other)
Collaborators: Aseer Central Hospital (Other Government); Khamis Mushayt General Hospital (Other Government)
Responsible Party: Principal Investigator, Snehil Dixit, Assistant Professor , Department of Medical Rehabilitation, King Khalid University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECM#2019-27
Record Dates: First submitted 2019-05-26; First posted 2019-09-03 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Following randomization, subjects will be assigned either to receive Intervention OR CONTROL (Standard Care) throughout the entire study period (parallel design)
Who Masked: Outcomes Assessor
Masking Description: An employee outside the research team will feed data into the computer in separate datasheets so that the researchers can analyze data without having access to information about the allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unsupported Upper extremity exercise (Active Comparator): Specially designed unsupported Arm exercises will be done for the population with a rating of somewhat hard 13-14 (Original scale) will be used as a guideline for intensity
  Interventions: Other: exercise
- Lower extremity exercise (Active Comparator): Specially designed Lower extremity exercises will be done for the population with a rating of somewhat hard 13-14 (Original scale) will be used as a guideline for intensity
  Interventions: Other: exercise
- Control (No Intervention): Here no active intervention will be given only standard care as prescribed by the hospital will be given

INTERVENTIONS:
Other: exercise — Stretching exercise for warmup, All arm exercise with and without weights as tolerated by the patients. Similarly lower limb exercise in different positions like lying standing as tolerated by the patients
  Arms: Lower extremity exercise; Unsupported Upper extremity exercise

SUMMARY:
Objective: is to find out the effect of unsupported upper extremity exercise versus lower extremity exercise on dyspnea and lung function

Methodology:

Sample and design: 60 patients with Randomized study design will be included in three groups.

Duration of intervention: Treatment will continue for 4 weeks. Outcome: Borgs scale and Medical Research Council scale (MRC) for dyspnea will be used to quantify the dyspnea. Lung function tests measure by PEFR, chronic obstructive pulmonary disease assessment test (CAT) will be used pre-post.

Discussion: We will compare three groups (UPPER EXTREMITY EXCERCISE (UEx), LOWER EXTREMITY EXERCISE (LEx), CONTROL (CON)) with COPD using interventional exercises for upper and lower extremities randomly assigned to three groups on the dyspnea symptoms and quantify and grade them pre-post the intervention. We will also use the CAT questionnaire pre-post to measure the changes in symptoms and functions.

DETAILED DESCRIPTION:
Background: Chronic Obstructive Pulmonary Disease (COPD) is one of the most common respiratory disorder affecting middle age group with progressing of symptoms worsening over time. The respiratory symptoms are persistent with compromised airflow due to small airway disorders or parenchymal abnormalities. The morbidity rate of COPD is about 251 million cases and mortality of 3.17 million per year globally with expected inflation in the future. The disease and death rate are well associated with dysfunction of skeletal muscle and cachexia. The amount of reduction in muscle strength of limbs is directly proportional to the severity of the disease. Dyspnea and decrement in endurance capacity will negatively affect the functional capability and quality of life in people suffering from COPD. Unsupported upper limb endurance training and lower limb endurance training showed significant improvement in Six-minute walk test and Quality of life.

Purpose: To determine the effect of Unsupported upper extremity endurance training and Unsupported lower extremity endurance training on dyspnea, lung function and quality of life.

Methodology: Study design: Randomized study design Study population: The people suffering from COPD referred by pulmonologist will be contacted for consent after oral explanation and answering all questions. After all the informed consents had been collected, randomization will be performed. The participants are randomly allocated to the Unsupported upper extremity endurance training (Experimental group-1), Unsupported lower extremity endurance training (Experimental group-2) and Conventional (Control group) prior to the first baseline assessment. The intensity of Exercise will be checked by the Original Borgs scale and Medical Research Council scale (MRC) for dyspnea.

Outcome measures: Lung function tests measures using PEFR, Airway Questionnaire 20 pre-post to measure the changes in symptoms and functions

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of COPD
* COPD secondary to any disease
* Age 10-70 years
* COPD in any stage according to GOLD classification

Exclusion Criteria:

* Taking any other form of alternative therapies
* The neurological deficit with the inability to understand of following instructions
* Recent Cardiovascular surgery patients
* Unstable angina patients
* Patients with musculoskeletal deficits

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-04-27 (Estimated)

PRIMARY OUTCOMES:
Airway Questionnaire 20 | Change is being evaluated from Baseline and at 4 wk
  The Airway Questionnaire 20 (AQ20) was developed for patients with asthma and chronic obstructive pulmonary disease (COPD). It contains 20 items, with scores ranging from 0 to 20 - high scores indicate poor QOL. It takes only a few minutes to complete and has been validated in asthma and COPD patients.
Borg's scale and Medical Research Council scale (MRC) for dyspnea | Change is being evaluated from Baseline and at 4 wk
  The Borg Rating of Perceived Exertion (RPE) scale will help you estimate how hard you're working (your activity intensity). Perceived exertion is how hard you think your body is exercising. Ratings on this scale are related to heart rate (how hard your heart is working to move blood through your body). Scale Range 6-20.
  Medical Research Council Scale of Breathlessness : The MRC breathlessness scale comprises five statements that describe almost the entire range of respiratory disability from none (Grade 1) to almost complete incapacity (Grade 5). It can be self-administered by asking subjects to choose a phrase that best describes their condition, e.g. 'I only get breathless with strenuous exertion' (Grade 1) or 'I am too breathless to leave the house' (Grade 5).

SECONDARY OUTCOMES:
Peak Expiratory Flow Rates (PEFR) | Change is being evaluated from Baseline and at 4 wk
  Peak expiratory flow rates, 80 to 100 percent of persons usual or "normal" peak flow rate signals all clear. 50 to 80 percent of persons or "normal" peak flow rate signals caution, Less than 50 percent of your usual or "normal" peak flow rate signals Medical alert.

CONTACTS AND LOCATIONS:
Locations (1):
- Snehil Dixit, Abhā, 'Asir Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
As we don't directly control the data. The data privacy is subjected to countries law and regulations